CLINICAL TRIAL: NCT06229470
Title: A Prospective, Multicenter, Single-arm Study Evaluating the Clinical Utility of Neurophysiological Measurements of ECAP-controlled Closed-loop Spinal Cord Stimulation (SCS) to Guide Treatment of Patients With Chronic Pain of the Trunk and/or Limbs.
Brief Title: Clinical Utility of Neurophysiological Measurements of ECAP-controlled Closed-loop SCS to Guide Treatment of Chronic Pain
Acronym: Neural Panel
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saluda Medical Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D103977
Record Dates: First submitted 2024-01-11; First posted 2024-01-29 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — Spinal Cord Stimulation; Drug Delivery Systems

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- ECAP-Controlled, Closed-Loop SCS (Experimental): Spinal cord stimulation that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude.
  Interventions: Device: Evoke Spinal Cord Stimulation (SCS) System

INTERVENTIONS:
Device: Evoke Spinal Cord Stimulation (SCS) System — A spinal cord stimulation (SCS) system that measures and records evoked compound action potentials (ECAPs) and automatically adjusts the stimulation current to maintain a consistent ECAP amplitude.

SUMMARY:
The purpose of this study is to evaluate the clinical utility of neurophysiological measurements of ECAP-controlled closed-loop SCS (i.e., neural panel metrics) to guide treatment of chronic pain of the trunk and/or limbs.

ELIGIBILITY:
Inclusion Criteria:

* Subject is planning to have a temporary trial with the Evoke System to aid in the management of chronic intractable pain of the trunk and/or limbs, including unilateral or bilateral pain associated with failed back surgery syndrome and/or intractable low back pain and leg pain.
* Leg pain score ≥ 6 cm (Visual Analog Scale [VAS]).
* Back pain score ≥ 6 cm (VAS).
* Subject is able to speak, read, and/or understand English, willing and capable of giving informed consent, and able to comply with study-related requirements, procedures, and visits.
* Subject is not pregnant and not <18 years of age.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Evoked Compound Action Potentials (ECAPs) as measured by the Evoke SCS System | through 6-months post-implant
  physiological parameter to be measured = Evoked Compound Action Potentials (ECAPs); measurement tool = Evoke SCS System

SECONDARY OUTCOMES:
Change in Visual Analogue Scale (VAS) Pain | through 6-months post-implant
  Visual Analogue Scale (VAS) to rate pain intensity (0mm [no pain] to 100mm [worst pain imaginable])
Change in PROMIS-29+2 | through 6-months post-implant
  PROMIS-29 Profile and 2 PROMIS Cognitive Function Abilities items. The PROMIS-29 is a 29-item profile instrument that assesses 8 universal domains (not disease-specific): Physical Function, Anxiety, Depression, Fatigue, Sleep Disturbance, Ability to Participate in Social Roles and Activities, Pain Interference, and Pain Intensity.
Change in PROMIS-10 Global Health | through 6-months post-implant
  10-item instrument that assesses Physical Health and Mental Health

CONTACTS AND LOCATIONS:
Locations (25):
- United States (25):
  - Lakeside Spine and Pain, Lake Havasu City, Arizona
  - Spanish Hills Interventional Pain Specialists, Camarillo, California
  - Pain Consultants of San Diego, La Mesa, California
  - Pacific Research Institute, Santa Rosa, California
  - Boomerang Healthcare, Walnut Creek, California
  - DBPS Research, Greenwood Village, Colorado
  - Pohlman Pain Associates, Delray Beach, Florida
  - Horizon Clinical Research, Jasper, Georgia
  - Rockford Pain Center, Rockford, Illinois
  - Goodman Campbell Brain and Spine, Carmel, Indiana
  - Metro Anesthesia & Pain Management, Des Moines, Iowa
  - Restorative Pain Institute, Louisville, Kentucky
  - Advanced Pain Institute, Hammond, Louisiana
  - Spine and Joint Institute, Glen Burnie, Maryland
  - Michigan Pain Specialists, Ann Arbor, Michigan
  - Pain Clinic of Michigan, Rochester Hills, Michigan
  - Tricity Research Center, LLC, Grand Island, Nebraska
  - Reno Tahoe Pain Associates, Reno, Nevada
  - Garden State Pain and Orthopedics, Clifton, New Jersey
  - Seaside Clinical Research Institute, Wilmington, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Premier Pain Treatment Institute, Loveland, Ohio
  - Carolinas Center for Advanced Management of Pain, Greenville, South Carolina
  - Institute of Precision Pain Medicine, Corpus Christi, Texas
  - Victoria Pain and Rehabilitation Center, Victoria, Texas

IPD SHARING:
Plan to Share IPD: No